CLINICAL TRIAL: NCT00278135
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of DHA on Cognitive Functions in the Elderly
Brief Title: Memory Improvement With Docosahexaenoic Acid Study (MIDAS)
Acronym: MIDAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005.1002
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Age-Related Cognitive Decline; Age-Related Memory Disorders
Keywords: Cognition; Memory; Nutrition; Omega-3; DHA
MeSH Terms: conditions — Memory Disorders | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: DHA (nutritional supplement) or placebo
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: DHA (nutritional supplement) or placebo

INTERVENTIONS:
Dietary Supplement: DHA (nutritional supplement) or placebo — oral 900mg/day

SUMMARY:
The purpose of this study is to investigate the effect of docosahexaenoic acid (DHA, 22:6n-3) in improving cognitive functions in subjects with age-related cognitive decline. DHA is a long chain omega-3 fatty acid (LC-PUFA) that plays an important role in neural and visual development and cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged 55 or greater.
* Have a subjective memory complaint and have a Logical Memory subtest (of the Wechsler Memory Scale - III [WMS-III]) raw score one standard deviation or greater below the mean of a younger population.
* Have the ability to understand the requirements of the study; be willing to provide written informed consent; and agree to abide by the study restrictions and return for the required assessments.
* If taking non-prohibited medication, be on a stable drug regimen (in prior 3 months).

Exclusion Criteria:

* Have a screening Mini-Mental State Examination (MMSE) < 26.
* Consume greater than 200 mg/day DHA as assessed on a DHA Food Frequency Questionnaire in the prior 2 months to screening.
* Use nutritional fish oil, flaxseed oil, omega-3 supplements, or huperzine in the prior 2 months to screening.
* Use acetylcholinesterase inhibitors or memantine in the prior 2 months to screening.
* Use major anti-psychotics or major anti-depressants.
* Use lipase inhibitors such as Xenical® (orlistat).
* History of major medical conditions including ischemic stroke, head trauma with loss of consciousness, epilepsy, psychosis, vascular dementia, depression (Geriatric Depression [15-item] > 5), myocardial infarction (within 1 year), uncontrolled diabetes, or blindness.
* History of major surgery within the past 6 months.
* Current use or history of drug and/or alcohol abuse within 5 years.
* Administration of any investigational product within the past 30 days.
* Inability to swallow capsules.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2005-12; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Determine the effects of DHA, a nutritional supplement (900 mg/d) on improving cognitive functions (i.e. working memory, memory retention, attention, and executive function) in healthy elderly subjects at 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Effects of DHA on visual acuity, levels of plasma phospholipids, and evaluating the safety and tolerability of the DHA dose administered | 24 weeks
The study will include a screening period, baseline, and 24 week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Yurko-Mauro, PhD, Study Director — DSM Nutritional Products, Inc.
Locations (14):
- United States (14):
  - Pivotal Research Center, Mesa, Arizona
  - Pacific Research Network, San Diego, California
  - Pacific Research Network, Vista, California
  - Radiant Research Denver, Denver, Colorado
  - Bradenton Neurology, Bradenton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Meridien Research, St. Petersburg, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Radiant Research Chicago, Chicago, Illinois
  - Clinical Trial Center, Jenkintown, Pennsylvania
  - Senior Adults Specialty Research, Austin, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - Radiant Research Salt Lake City, Salt Lake City, Utah
  - Neurological Research Center, Inc., Bennington, Vermont

REFERENCES:
- [Derived] Yurko-Mauro K, McCarthy D, Rom D, Nelson EB, Ryan AS, Blackwell A, Salem N Jr, Stedman M; MIDAS Investigators. Beneficial effects of docosahexaenoic acid on cognition in age-related cognitive decline. Alzheimers Dement. 2010 Nov;6(6):456-64. doi: 10.1016/j.jalz.2010.01.013. PMID 20434961